CLINICAL TRIAL: NCT06905080
Title: Dialysis Catheter Caps Case Feasibility Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephanie R. Jenkins, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 24-010774
Record Dates: First submitted 2025-03-18; First posted 2025-04-01 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Sterile Catheter; Catheter-related Bloodstream Infections; Dialysis Catheter; Dialysis
Keywords: Sterile Catheter; catheter-related bloodstream infections; Catheter Caps Case; infection control; C3; Dialysis Catheter Caps Case; Dialysis Catheter; Dialysis; Catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Catheter Caps Case (C3) — The nursing team will then assess the participant's catheter, catheter site, and lumens. The C3 device will be placed on the distal lumens and hub caps of the participant's hemodialysis catheter using clean technique and left in place for approximately 15 minutes. During this time, the participant will be asked to lay, sit, and stand while wearing the C3 device. The RN will stay with the participant during the entire time and will write down any comments or requests regarding the C3 made by the participant. After 15 minutes, the nursing team will remove the C3 device and reassess the condition of the catheter site and lumens, noting any changes. Finally, the participant will complete a 10 item post- intervention survey, developed by the study team and evaluated for face validity by all members of the team to provide feedback on the design of the C3 device.

SUMMARY:
The purpose of this research is to evaluate patient comfort and ease of an investigational device called Catheter Caps Case (C3) attached to the hemodialysis catheter over a 15-minute period. You have been asked to take part in this research because you have been identified as a dialysis patient with a hemodialysis catheter.

DETAILED DESCRIPTION:
Tunneled hemodialysis catheters are commonly used to administer dialysis to patients with kidney failure to remove excess fluid and waste from the blood. Traditionally, the maintenance and protection of these catheters involves the use of gauze and tape to secure the catheter and cover the double lumen and caps. While this method is widely practiced, it has several drawbacks that can affect both patient outcomes and healthcare efficiency.

Firstly, the use of gauze and tape can be uncomfortable for patients. The adhesive nature of the tape can cause skin irritation and allergic reactions, in addition the gauze can impede visualization of the entire length of the catheter. Additionally, the process of routine changing gauze and tape is time-consuming for healthcare providers and can increase the risk of catheter dislodgment during or catheter caps disconnection during removal of tape gauze combination.

Another significant concern is infection control. Gauze and tape do not provide an optimal sterile barrier, which can lead to an increased risk of catheter-related bloodstream infections (CRBSIs). These infections are associated with prolonged hospital stays, higher hospital healthcare costs, and increased patient mobility and mortality.

The catheter caps case was developed to address these issues by providing a more secure and sterile alternative to gauze and tape. The case is designed to cover the catheter's double lumen and end caps, offering added protection and stability. Its innovative design aims to reduce the risk of accidental dislodgement, enhance infection control, and improve overall patient comfort by eliminating the need for gauze and adhesive tape.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with tunneled dialysis catheter that will not be removed in the next 90 days.
2. Patients from the home dialysis program or in-center (outpatient dialysis) patient population.
3. Patients who are age 18 years or older

Exclusion Criteria:

1. Patient-delayed graft function (DGF)
2. Acute kidney injury patients
3. Patients with non-tunneled catheter
4. Allergies to the BioMed Elastic 50A Resin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the ease and structural integrity of the Catheter Caps Case (C3) | 1 Day
  The feasibility of the catheter cap will be assessed by evaluating its ease of use and structural integrity. This includes measuring the time required for secure placement and removal compared to traditional gauze and tape, as well as obtaining standardized usability ratings from healthcare providers. Additionally, the study will track the incidence of accidental catheter dislodgement during routine cap changes to determine whether the cap provides enhanced stability.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic (Florida), Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this time, it has not been determined whether individual participant data (IPD) will be shared. The decision will depend on factors such as regulatory requirements, ethical considerations, and sponsor policies. If IPD sharing is implemented, appropriate safeguards will be in place to protect participant confidentiality.